CLINICAL TRIAL: NCT05324384
Title: Different Doses of Sirolimus for the Maintenance Treatment of Kaposiform Hemangioendothelioma: a Randomized Controlled Trial
Brief Title: Different Doses of Sirolimus for the Maintenance Treatment of Kaposiform Hemangioendothelioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Principal Investigator, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-405
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Hemangioendothelioma
Keywords: Kaposiform hemangioendothelioma; Hemangioendothelioma; Sirolimus
MeSH Terms: conditions — Hemangioendothelioma; Kaposiform Hemangioendothelioma | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose of sirolimus (Experimental): The plasma trough concentration of sirolimus is maintained within the range of 10-15 ng/ml by adjusting sirolimus dose, for 6 months. Then, The plasma trough concentration of sirolimus is maintained within the range of 5-8 ng/ml by adjusting sirolimus dose, for 6 months.
  Interventions: Drug: Sirolimus
- Regular dose of sirolimus (Active Comparator): Sirolimus The plasma trough concentration of sirolimus is maintained within the range of 10-15 ng/ml by adjusting sirolimus dose, for 1 year.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Use of different doses of the same drug
  Other Names: Rapamycin; Rapamune

SUMMARY:
The purpose of this study is to compare the efficacy and safety of different doses of sirolimus in the maintenance treatment of kaposiform hemangioendothelioma.

DETAILED DESCRIPTION:
Kaposiform hemangioendothelioma (KHE) is a rare aggressive vascular neoplasm that occurs predominantly in infancy or early childhood, with an incidence of approximately 0.071/100,000. Currently, sirolimus is a promising treatment modality for KHE. Most scholars consider sirolimus blood concentration of 5-15 ng/ml to be an effective therapeutic concentration, while 10-15 ng/ml is the most commonly used blood concentration. However, long-term higher dose sirolimus treatment can cause some common adverse effects, such as oral mucositis which affects the quality of life of the patient. Finer control of the plasma concentration of sirolimus may contribute to the efficacy of treatment and reduce the incidence of complications. Previous studies have found good efficacy of low-dose sirolimus maintenance treatment for KHE. However, there is no high-level evidence to support this treatment strategy. Therefore, we conducted this study to find out whether an early reduction in sirolimus dose would benefit the prognosis of the patients.

ELIGIBILITY:
Inclusion Criteria:

Presenting a KHE with the following characteristics:

1. Male and female;
2. Between 0 and 14 years of age;
3. Diagnosis of KHE as determined by:

   * Biopsy;
   * Compatible MRI findings;
   * History and clinical features.
4. Patients were required to have adequate liver, renal and bone marrow function, and absence of active infection
5. Consent of parents (or the person with parental authority in families): signed and dated written informed consent.

Exclusion Criteria:

1. Patients contraindicated for the administration of sirolimus (e.g., those with an allergy to sirolimus or other rapamycin analog)
2. Exposure to chemotherapy, embolization, corticosteroids, propranolol, sclerotherapy or any other investigational agents within 1 weeks before enrolment on study;
3. Patients had a history of a major surgery within 2 weeks before enrollment;
4. Patients who have a history of treatment with sirolimus or other mTOR inhibitor;
5. Any known evidence of significant local or systemic uncontrolled infection, defined as receiving intravenous antibiotics at the time of enrollment;
6. Concurrent severe and/or uncontrolled medical diseases that could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe malnutrition, chronic liver or renal disease, active upper gastrointestinal tract ulceration).
7. Impairment of gastrointestinal function or chronic gastrointestinal disease that may significantly alter the absorption of sirolimus.
8. Patients with inadequate liver function:

   Total bilirubin higher than or equal to 1.5 × the upper limit of the normal (ULN) for age and alanine aminotransferase and aspartate aminotransferase higher than or equal to 2.5 × the ULN for age.
9. Patients with inadequate renal function:

   0-5 years of age maximum serum creatinine (mg/dL) of 0.8; 6-10 years of age maximum serum creatinine (mg/dL) of 1.0; 11-14 years of age maximum serum creatinine (mg/dL) of 1.2;
10. Adequate bone marrow function:

    Absolute neutrophil count lower than 1 × 109/L;
11. History of a malignancy within 5 years;
12. HIV infection or known immunodeficiency;
13. Indication for treatment with corticosteroids, vincristine, interferon-α, sirolimus, or tacrolimus for an indication other than IH;
14. Patients with an inability to participate in or follow-up during the study treatment and assessment plan;
15. Inability to give informed consent.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The changes in KHE volume | 12 months.
  Response to therapy was measured by volumetric magnetic resonance imaging (MRI) analyses were performed at baseline and 6 and 12 months after treatment and were independently assessed by 2 radiologists. Changes in KHE size were classified as further growth (increase of ≥10%), no change (<10% increase and <10% decrease), partial involution (decrease of ≥10% and <75%), nearly complete involution (decrease of ≥75% and <100%), or complete involution (100%).

SECONDARY OUTCOMES:
Quality of life (QOL) in patients | Baseline, 6 months, 12 months.
  Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Genetic Core Infant Scales (<2 years) or Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Genetic Core Scales (2-18 years) were used.
Frequency of adverse events | Baseline, 6 months, 12 months.
  Frequency of adverse events (e.g. gastrointestinal disorders, blood and lymphatic system disorders, metabolic disorders or other abnormal laboratory results, skin disorders and general disorders, etc.) collected by investigator and reported by parents. All adverse events were collected and graded according to Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE v4.0). The causality of the adverse event was determined by the multidisciplinary staff and was classified as definitively not related, probably not related, possibly related, probably related, or definitively related. Any dose reductions, interruptions, or cessations enacted at the discretion of the investigators were recorded.
The changes in the patient's musculoskeletal complication. | Baseline, 3 monthss, 6 months, 9 months, 12 months.
  The severity of musculoskeletal complication was scored by using a 4-point scale: 1, asymptomatic or mild symptoms, clinical or diagnostic observations only; 2, moderate symptoms, limiting age-appropriate instrumental activities of daily living; 3, severe or medically significant symptoms, disabling or limiting self-care activities of daily living; and 4, life-threatening consequences, with urgent intervention indicated.
The changes of platelet counts. | Baseline, 3 monthss, 6 months, 9 months, 12 months.
  Platelet counts
The changes of fibrinogen levels. | Baseline, 3 monthss, 6 months, 9 months, 12 months.
  Fibrinogen levels
The changes of D-dimer levels. | Baseline, 3 monthss, 6 months, 9 months, 12 months.
  D-dimer levels

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, MD, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ji Y, Chen S, Yang K, Xia C, Li L. Kaposiform hemangioendothelioma: current knowledge and future perspectives. Orphanet J Rare Dis. 2020 Feb 3;15(1):39. doi: 10.1186/s13023-020-1320-1. PMID 32014025
- [Result] Wang Z, Yao W, Sun H, Dong K, Ma Y, Chen L, Zheng S, Li K. Sirolimus therapy for kaposiform hemangioendothelioma with long-term follow-up. J Dermatol. 2019 Nov;46(11):956-961. doi: 10.1111/1346-8138.15076. Epub 2019 Sep 5. PMID 31489702
- [Result] Ji Y, Chen S, Xiang B, Li K, Xu Z, Yao W, Lu G, Liu X, Xia C, Wang Q, Li Y, Wang C, Yang K, Yang G, Tang X, Xu T, Wu H. Sirolimus for the treatment of progressive kaposiform hemangioendothelioma: A multicenter retrospective study. Int J Cancer. 2017 Aug 15;141(4):848-855. doi: 10.1002/ijc.30775. Epub 2017 May 26. PMID 28486787
- [Result] Croteau SE, Liang MG, Kozakewich HP, Alomari AI, Fishman SJ, Mulliken JB, Trenor CC 3rd. Kaposiform hemangioendothelioma: atypical features and risks of Kasabach-Merritt phenomenon in 107 referrals. J Pediatr. 2013 Jan;162(1):142-7. doi: 10.1016/j.jpeds.2012.06.044. Epub 2012 Aug 4. PMID 22871490
- [Result] Rossler J, Baselga E, Davila V, Celis V, Diociaiuti A, El Hachem M, Mestre S, Haeberli D, Prokop A, Hanke C, Loichinger W, Quere I, Baumgartner I, Niemeyer CM, Kapp FG. Severe adverse events during sirolimus "off-label" therapy for vascular anomalies. Pediatr Blood Cancer. 2021 Aug;68(8):e28936. doi: 10.1002/pbc.28936. Epub 2021 Feb 13. PMID 33580918
- [Result] Ji Y, Chen S, Zhou J, Yang K, Zhang X, Xiang B, Qiu T, Gong X, Zhang Z, Lan Y, Hu F, Kong F, Qiu Q, Zhang Y. Sirolimus plus prednisolone vs sirolimus monotherapy for kaposiform hemangioendothelioma: a randomized clinical trial. Blood. 2022 Mar 17;139(11):1619-1630. doi: 10.1182/blood.2021014027. PMID 35030255